CLINICAL TRIAL: NCT07065266
Title: The Utility of a Dichotomous Pain Scale in Reducing Postoperative Opioids Consumption in Outpatient ACL Surgery: A Prospective Randomized Controlled Study
Brief Title: Does the Use of a Simplified Pain Questionnaire Impact Opioid Consumption Among People Receiving Anterior Cruciate Ligament (ACL) Knee Surgery?
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Todd Alamin, Professor of Orthopaedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 45010
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Anterior Cruciate Ligament (ACL) Reconstruction; Anterior Cruciate Ligament/Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-point pain scale (Active Comparator): participants undergoing ACL reconstructive surgery are asked to use a 10-point NPRS pain scale to describe their pain post-operatively
  Interventions: Other: Numerical Pain Rating Scale (NPRS)
- Binary pain questionnaire (Experimental): Participants undergoing ACL reconstructive surgery are asked to describe their pain as tolerable or intolerable post-operatively
  Interventions: Other: Binary pain questionnaire

INTERVENTIONS:
Other: Binary pain questionnaire — Post-operative questionnaire that asks if pain is 'tolerable' or 'intolerable'
  Arms: Binary pain questionnaire
Other: Numerical Pain Rating Scale (NPRS) — Standard 10-point pain scale used post-operatively to assess pain
  Arms: 10-point pain scale

SUMMARY:
The goal of this randomized clinical trial is to compare opioid consumption among patients who receive a binary pain scale compared to those who receive a standard 10-point pain scale after undergoing anterior cruciate ligament (ACL) reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Undergoing ACL reconstruction surgery at Stanford Sports Medicine Redwood City, with autograft or allograft, with or without concomitant meniscal repair.

Exclusion Criteria:

* Pregnant women
* Surgical history of the operated knee
* Known allergy to opioid medications
* Received extra-routine pain care (as compared with the average ACL patients at the Sports Medicine division) given by the anesthesiologists, such as the postoperative epidural analgesia or the ultra-sound guided femoral nerve block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Amount of opioid medication used post-operatively for 14 days | 14 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Todd Alamin, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Orthopaedic and Sports Medicine, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No